CLINICAL TRIAL: NCT03258827
Title: Chang Gung Medical Hospital
Brief Title: Outcome of Exercise With a Towel in Elderly With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201700238B0
Record Dates: First submitted 2017-07-18; First posted 2017-08-23 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-07

CONDITIONS: Sarcopenia
Keywords: elderly; sarcopenia; strengthening exercise
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: We randomize these 60 older adults into 2 groups (experimental group and control group) and there are 30 older adults in each group. Those older adults are age above 65 year-old, have lower grip strength and slower walking speed. Experimental group receive this exercise program training, 60 minutes/time, 3 times/week, total duration: 3 months. Home-based program focuses on walking activity at fast speed, 3 times/week, 60 minutes/times, would be assigned for Control group. Total duration is 3 months.
Who Masked: Outcomes Assessor
Masking Description: The assistant who doesn't know the group which patients belong to will evaluate the functional performance of the patients three times, such as before training, after training, post-training 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with a towel (Experimental): There are 30 old adults in this group who receives exercise program with a towel.
  Interventions: Procedure: Exercise with a towel
- Home-based exercise (Placebo Comparator): There are 30 old adults in this group who is suggested a home-based program focuses on walking activity at fast speed.
  Interventions: Procedure: Home-based exercise

INTERVENTIONS:
Procedure: Exercise with a towel — Exercise program composes with warm-up, strengthening exercise, cold-down, 60 minutes/time, 3 times/week. A towel is an important tool for exercise. Total duration of the program is 3 months.
  Other Names: Home-based exercise
  Arms: Exercise with a towel
Procedure: Home-based exercise — Home-based program focuses on walking activity at fast speed, 3 times/week, 60 minutes/times. The total duration is 3 months.
  Arms: Home-based exercise

SUMMARY:
As the proportion of older adults increases, elderly-related issues attract more attention. Sarcopenia is one of the popular elderly-related issues. Sarcopenia may induce decreased muscle strength, poor physical activity, even disability and increase rate of hospitalization and mortality. Therefore, we want to figure out the management for decreasing prevalence of sarcopenia in older adults. This trial is planned to perform during 2017/08/01~2017/12/31. We plan to enroll 60 elderlies who are sarcopenia. These patient will be divided into 2 group randomize. Experimental group will be received a set of exercise, composed by warm-up, strengthening training with a towel, cold-down, 60 minutes per time, 3 times per week. Control group will be suggested home-based walking activity. We will evaluate the patient's functional performance three times, before training, after training, post-training for three months, respectively. These results will be analyzed by repeated measure ANOVA.

DETAILED DESCRIPTION:
As the proportion of older adults increases, elderly-related issues attract more attention. Sarcopenia is one of the popular elderly-related issues. Skeletal muscle is an important component for sustaining physical activity and storing protein. Protein of skeletal muscle is used as energy substrates in cases of starvation or under stress. As being aging, physical condition degenerates gradually. Older adults usually have multiple chronic diseases. Lesser physical function results in less physical activity. As a result, more muscle mass would be lost. In previous study, after the age of 50 year-old, muscle mass decreases 1-2% per year. The velocity of muscle mass decline increases after the age of 60 year-old. Sarcopenia may induce decreased muscle strength, poor physical activity, even disability and increase rate of hospitalization and mortality. Therefore, we want to figure out the management for decreasing prevalence of sarcopenia in older adults.

Exercise is an important method for preventing sarcopenia. In this study, we intend to design a set of exercise which is easily performed for older adults and also has preventing muscle mass loss effect. Towel is an important tool for exercise.

Duration to execute is during 2017/08/01~2017/12/31. We randomize these 60 older adults into 2 groups (experimental group and control group) and there are 30 older adults in each group. Those older adults are age above 65 year-old, have lower grip strength and slower walking speed. One assistant who doesn't know which group these older adults belonged to would record their basic information and is responsible for the evaluation. We will evaluate the older adults' functional performance three times, before training, after training, post-training for three months, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. age above 65 y/o
2. low muscle mass (male<7.0 kg/m2, female<5.4kg/m2, tested by Dual energy X-ray Absorptiometry)
3. with or without low grip strength (male< 26 kg, female <18 kg)
4. with or without low walk speed (≤ 0.8 m/s).

Exclusion Criteria:

1. cognitive impairment or can't follow order appropriately
2. elderlies with medical problems that they can't perform the exercise program

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Fat mass | Baseline
  Dual-energy X-ray absorptiometry is used for measuring fat mass.
Fat-free mass | Baseline
  Dual-energy X-ray absorptiometry is used for measuring fat-free mass.
Bone mineral density | Baseline
  Dual-energy X-ray absorptiometry is used for measuring bone mineral density.
Maximal grip strength | Baseline
  Handgrip dynamometer is used for measuring maximal grip strength.
Walking speed | Baseline
  Participants are asked to walk at a comfortable speed to perform 10 meter walk test.
Timed up and go test | Baseline
  At first, the participant sits down. Then the participant would be asked to stand up, walk straight for 3 meters, turn around, go back to the chair and sit down. The duration of whole test would be measured.
Times of stand-up and sit-down within 30 seconds | Baseline
  The participant is asked to cross arm before the chest. The investigator would record the times of stand-up and sit-down within 30 seconds.
6 minutes walking test | Baseline
  At first, the participant sits down for a rest for 10 minutes. The participant would be asked to walk as longer distance as the participant can within 6 minutes.
Berg balance test | Baseline
  The investigator record scores of 14 items involved in Berg balance test for measuring balance of the old adults.

SECONDARY OUTCOMES:
Fat mass | Change between baseline and 3 month after training
  Dual-energy X-ray absorptiometry is used for measuring fat mass
Fat mass | Change between baseline and 6 month after training
  Dual-energy X-ray absorptiometry is used for measuring fat mass
Fat-free mass | Change between baseline and 3 month after training
  Dual-energy X-ray absorptiometry is used for measuring fat-free mass
Fat-free mass | Change between baseline and 6 month after training
  Dual-energy X-ray absorptiometry is used for measuring fat-free mass
Bone mineral density | Change between baseline and 3 month after training
  Dual-energy X-ray absorptiometry is used for measuring bone mineral density
Bone mineral density | Change between baseline and 6 month after training
  Dual-energy X-ray absorptiometry is used for measuring bone mineral density
Maximal grip strength | Change between baseline and 3 month after training
  Handgrip dynamometer is used for measuring maximal grip strength.
Maximal grip strength | Change between baseline and 6 month after training
  Handgrip dynamometer is used for measuring maximal grip strength.
Walking speed | Change between baseline and 3 month after training
  Participants are asked to walk at a comfortable speed to perform 10 meter walk test.
Walking speed | Change between baseline and 6 month after training
  Participants are asked to walk at a comfortable speed to perform 10 meter walk test.
Timed up and go test | Change between baseline and 3 month after training
  At first, the participant sits down. Then the participant would be asked to stand up, walk straight for 3 meters, turn around, go back to the chair and sit down. The duration of whole test would be measured.
Timed up and go test | Change between baseline and 6 month after training
  At first, the participant sits down. Then the participant would be asked to stand up, walk straight for 3 meters, turn around, go back to the chair and sit down. The duration of whole test would be measured.
Times of stand-up and sit-down within 30 seconds | Change between baseline and 3 month after training
  The participant is asked to cross arm before the chest. The investigator would record the times of stand-up and sitdown within 30 seconds.
Times of stand-up and sit-down within 30 seconds | Change between baseline and 6 month after training
  The participant is asked to cross arm before the chest. The investigator would record the times of stand-up and sitdown within 30 seconds.
6 minutes walking test | Change between baseline and 3 month after training
  At first, the participant sits down for a rest for 10 minutes. The participant would be asked to walk as longer distance as the participant can within 6 minutes.
6 minutes walking test | Change between baseline and 6 month after training
  At first, the participant sits down for a rest for 10 minutes. The participant would be asked to walk as longer distance as the participant can within 6 minutes.
Berg balance test | Change between baseline and 3 month after training
  The investigator record scores of 14 items involved in Berg balance test for measuring balance of the old adults.
Berg balance test | Change between baseline and 6 month after training
  The investigator record scores of 14 items involved in Berg balance test for measuring balance of the old adults.

CONTACTS AND LOCATIONS:
Overall Officials: Shui Tseng, Study Chair — Chang Gung Medical Foundation Institutional Review Board
Locations (1):
- Wujia Senior Citizens activity Center of Kaohsiung City Government, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No